CLINICAL TRIAL: NCT06701383
Title: Randomized Comparison Between 3 D CT Overlay and Conventional Fluoroscopy to Decrease Contrast and Radiation Exposure During Cryoballoon Ablation for Atrial Fibrillation
Acronym: CAFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety point reached, subjects in the 3D CT overlay group received sugnificantly less contrast.
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, B. Oude Velthuis, cardiologist, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL39065.044.11; P12-16 (Other: METC Twente)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard fluorscopy (Active Comparator): Cryoablation using a balloon with standard fluoroscopy
  Interventions: Device: Cryoablation
- 3D CT overlay (Experimental): Cryoablation using a balloon with 3D CT overlay
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Pulmonary vein isolation using cryoablation

SUMMARY:
Cryoablation using a balloon is an effective therapy for paroxysmal atrial fibrillation (AF), however associated with significant amounts of radiation exposure and contrast medium use. A new imaging technique (3D CT overlay) could reduce radiation exposure and contrast medium use significantly.

ELIGIBILITY:
Inclusion Criteria:

- All patients screened are accepted for PVI according to the current guidelines - Patients are candidates for enrolment if they have paroxysmal AF as defined in the guidelines

Exclusion Criteria:

* Persistent, long-standing persistent or permanent AF
* Left atrial diameter > 50 mm (measured in the parasternal long axis, as assessed with transthoracic echocardiography)
* Previous PVI ablation (epicardial or endocardial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy time | Procedure time
  To compare the fluoroscopy time between cryoballoon ablation with and without the use of 3D CT overlay
radiation exposure | Procedure time
  To compare the radiation exposure (DAP) between cryoballoon ablation with and without the use of 3D CT overlay
Contrast | Amount of contrast during procedure
  To compare the amount of contrast medium between cryoballoon ablation with and without the use of 3D CT overlay

SECONDARY OUTCOMES:
Recurrence | one year
  The percentage of patients without a recurrence of AF, without AADs, within a follow-up period of at least 12 months after a stabilisation period of 90 days after the initial procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jurren van Opstal, MD, PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands